CLINICAL TRIAL: NCT02752906
Title: Immunogenicity and Safety of a Booster Dose of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Adolescents and Adults
Brief Title: Immunogenicity and Safety of a Booster Dose of an Investigational Quadrivalent Meningococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MET56; U1111-1161-2710 (Other: WHO); 2018-001470-18 (EudraCT Number)
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; MenACYW Conjugate vaccine; Licensed Meningococcal Conjugate Vaccine (MCV4)
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal vaccine-primed adolescents (greater than or equal to [>=] 15 to less than [< ]18 years) or adults (>= 18 years) received a single dose of a MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Menactra® (Active Comparator): Healthy, meningococcal- vaccine-primed adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of Menactra ® vaccine on Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular
  Other Names: MenACYW Conjugate vaccine
  Arms: MenACYW Conjugate Vaccine
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra®

SUMMARY:
The aim of the study was to describe the safety and antibody response to booster administration with Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine in participants who received their first quadrivalent meningococcal Conjugate vaccine dose in the past 4-10 years.

Primary Objective:

* To demonstrate the non-inferiority of the vaccine seroresponse of meningococcal serogroups A, C, Y, and W following the administration of a booster dose of MenACYW Conjugate vaccine compared to those observed following the administration of a booster dose of Menactra® in participants who were first vaccinated with 1 dose of a quadrivalent meningococcal vaccine 4 to 10 years before the booster dose.

Secondary Objectives:

* To evaluate the vaccine seroresponse of meningococcal serogroups A, C, Y, and W measured using human serum bactericidal assay (hSBA) in serum specimens collected 6 days after vaccination in a subset of 120 participants.
* To evaluate the antibody responses (geometric mean titers) to serogroups A, C, Y, and W measured using hSBA on Day 0 (pre-vaccination) and Day 30 after vaccination.

Observational Objectives:

* To describe the antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA assessed at Day 0, Day 6, and Day 30 days after vaccination.
* To describe the antibody responses to the meningococcal serogroups A, C, Y, and W before and 30 days after vaccination with MenACYW Conjugate vaccine or Menactra® measured by rabbit serum bactericidal assay (rSBA) in a subset of participants.
* To describe the safety profile of MenACYW Conjugate vaccine compared to that of a licensed Menactra® after booster vaccination.

DETAILED DESCRIPTION:
Healthy adolescents and adults who had received 1 dose of a quadrivalent meningococcal Conjugate vaccine 4 to 10 years previously were randomized to receive either 1 dose of MenACYW Conjugate vaccine or licensed Menactra®. All participants underwent immunogenicity assessment at baseline (pre-vaccination) and post-vaccination and were also evaluated for safety up to Day 180 post-vaccination. In addition, a subset had an additional blood sample collected at 6 days post-vaccination for immunogenicity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 15 years on the day of inclusion.
* Participant has documented record of having received 1 dose of a quadrivalent meningococcal conjugate vaccine 4 to 10 years prior to study vaccination.
* Participant aged 15 to < 18 years: assent form signed and dated by the participant and informed consent form (ICF) signed and dated by the parent or guardian.
* Participant aged >=18 years: ICF signed and dated by the participant.
* Participants aged 15 to < 18 years: both the participant and parent / guardian were able to attend all scheduled visits and to comply with all trial procedures.
* Participants aged >= 18 years: able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine before Day 30 visit except for influenza vaccination, which may be received at least 2 weeks before study investigational vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either an investigational or approved meningococcal B vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Personal history of Guillain-Barré syndrome.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to the Investigator's judgment) on the day of vaccination or febrile illness (temperature >= 100.4°Fahrenheit [F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (30):
- United States (29):
  - Investigational Site Number 016, Birmingham, Alabama
  - Investigational Site Number 032, Dothan, Alabama
  - Investigational Site Number 026, Mesa, Arizona
  - Investigational Site Number 022, Jonesboro, Arkansas
  - Investigational Site Number 005, Downey, California
  - Investigational Site Number 014, La Puente, California
  - Investigational Site Number 029, San Diego, California
  - Investigational Site Number 001, San Diego, California
  - Investigational Site Number 013, Bardstown, Kentucky
  - Investigational Site Number 027, Nicholasville, Kentucky
  - Investigational Site Number 015, Metairie, Louisiana
  - Investigational Site Number 018, Woburn, Massachusetts
  - Investigational Site Number 010, Troy, Michigan
  - Investigational Site Number 008, Kansas City, Missouri
  - Investigational Site Number 028, St Louis, Missouri
  - Investigational Site Number 023, Lincoln, Nebraska
  - Investigational Site Number 031, Omaha, Nebraska
  - Investigational Site Number 006, Rochester, New York
  - Investigational Site Number 012, Fargo, North Dakota
  - Investigational Site Number 019, Cincinnati, Ohio
  - Investigational Site Number 011, Fairfield, Ohio
  - Investigational Site Number 025, Huber Heights, Ohio
  - Investigational Site Number 021, Kettering, Ohio
  - Investigational Site Number 009, Erie, Pennsylvania
  - Investigational Site Number 007, Hermitage, Pennsylvania
  - Investigational Site Number 024, Tullahoma, Tennessee
  - Investigational Site Number 020, Salt Lake City, Utah
  - Investigational Site Number 003, Salt Lake City, Utah
  - Investigational Site Number 017, South Jordan, Utah
- Investigational Site Number 030, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Anez G, Hedrick J, Simon MW, Christensen S, Jeanfreau R, Yau E, Pan J, Jordanov E, Dhingra MS. Immunogenicity and safety of a booster dose of a quadrivalent meningococcal tetanus toxoid-conjugate vaccine (MenACYW-TT) in adolescents and adults: a Phase III randomized study. Hum Vaccin Immunother. 2020 Jun 2;16(6):1292-1298. doi: 10.1080/21645515.2020.1733867. Epub 2020 Mar 25. PMID 32209015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 30 centers from 15 April 2016 to 02 August 2016.
Pre-assignment Details: A total of 810 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized in the study.
Groups:
- MenACYW Conjugate Vaccine: Healthy, meningococcal vaccine-primed adolescents (greater than or equal to [>=] 15 to less than [<] 18 years) or adults (>= 18 years) received a single dose of a Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine on Day 0.
- Menactra ®: Healthy, meningococcal-vaccine-primed adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra ®) vaccine on Day 0.
Period: Overall Study
Arm/Group | MenACYW Conjugate Vaccine | Menactra ®
Started | 403 | 407
Vaccinated | 402 | 407
Completed | 396 | 402
Not Completed | 7 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- MenACYW Conjugate Vaccine: Healthy, meningococcal vaccine-primed adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of a MenACYW Conjugate vaccine on Day 0.
- Menactra ®: Healthy, meningococcal-vaccine-primed adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of Menactra ® vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | MenACYW Conjugate Vaccine | Menactra ® | Total
Number analyzed (Participants) | 403 | 407 | 810
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (5.96) | 19.9 (5.59) | 20.0 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 200 | 407
  Male | 196 | 207 | 403
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 40 | 46 | 86
  White | 342 | 340 | 682
  More than one race | 8 | 17 | 25
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 403 | 407 | 810

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroresponse to Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine
Description: The serum bactericidal assay using human complement (hSBA) vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:16 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >= 1:8.
Time Frame: Day 30 (post-vaccination)
Population: Per-Protocol Analysis Set-2 (PPAS2): included all participants who had no protocol deviations (not meet inclusion/exclusion criteria, participant did not received vaccine, administration of vaccine not done as per-protocol). PPAS2 defined for evaluating the immune response of MenACYW vaccine measured by hSBA assessed at Day 30 after vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine | Menactra ®
Number analyzed (Participants) | 384 | 389
percentage of participants
  Serogroup A | 92.2 [89.0 to 94.7] | 87.1 [83.4 to 90.3]
  Serogroup C | 97.1 [94.9 to 98.6] | 91.8 [88.6 to 94.3]
  Serogroup Y | 97.4 [95.3 to 98.7] | 95.6 [93.1 to 97.4]
  Serogroup W | 98.2 [96.3 to 99.3] | 90.7 [87.4 to 93.4]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine vs Menactra ®; Serogroup A; Test type: Non-Inferiority — 95% confidence interval (CI) of the difference was calculated from the Wilson Score Method without continuity correction. If the lower limit of the 2-sided 95% CI of the difference between the 2 percentage was > -10%, the non- inferiority assumption was rejected; Percentage Difference = 5.0, 95% CI 2-sided [0.735 to 9.38]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine vs Menactra ®; Serogroup C; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. If the lower limit of the 2-sided 95% CI of the difference between the 2 percentage was > -10%, the non-inferiority assumption was rejected; Percentage Difference = 5.4, 95% CI 2-sided [2.16 to 8.76]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine vs Menactra ®; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 1.8, 95% CI 2-sided [-0.907 to 4.55]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine vs Menactra ®; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage Difference = 7.4, 95% CI 2-sided [4.30 to 10.9]

2. Secondary Outcome: Percentage of Participants With Seroresponse to Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine at Day 6 After Vaccination
Description: The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:16 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >= 1:8.
Time Frame: Day 6 (post-vaccination)
Population: Per-Protocol Analysis Set-1 (PPAS1): included all participants who received at least 1 dose of study vaccine(s) and had no protocol deviations (not meet inclusion/exclusion criteria, participant did not received vaccine). PPAS1 defined for evaluating the immune response of MenACYW vaccine measured by hSBA assessed at Day 6 after vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine | Menactra ®
Number analyzed (Participants) | 55 | 62
percentage of participants
  Serogroup A | 72.7 [59.0 to 83.9] | 66.1 [53.0 to 77.7]
  Serogroup C | 83.6 [71.2 to 92.2] | 87.1 [76.1 to 94.3]
  Serogroup Y | 90.9 [80.0 to 97.0] | 83.9 [72.3 to 92.0]
  Serogroup W | 94.5 [84.9 to 98.9] | 83.9 [72.3 to 92.0]

3. Secondary Outcome: Geometric Mean Titers Against Meningococcal Serogroups A, C, Y, and W Antibodies Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine
Description: Meningococcal antibody responses against Serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS2.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | MenACYW Conjugate Vaccine | Menactra ®
Number analyzed (Participants) | 384 | 389
titers (1/dilution)
  Serogroup A | 497 [436 to 568] | 296 [256 to 343]
  Serogroup C | 2618 [2227 to 3078] | 599 [504 to 711]
  Serogroup Y | 2070 [1807 to 2371] | 811 [699 to 941]
  Serogroup W | 1747 [1508 to 2025] | 723 [614 to 853]

4. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions or Systemic Reactions Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine
Description: A Solicited Reaction (SR) was an Adverse Event (AE) that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). Solicited injection site reactions: Pain (Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significantly prevent daily activity), erythema and swelling (Grade 1: >=25 millimeter [mm] to <= 50 mm, Grade 2: >=51 to <=100 mm, Grade 3: > 100 mm). Solicited systemic reactions: Fever (Grade 1: >=38.0 degree Celsius (°C) to <=38.4°C, Grade 2: >=38.5°C to <=38.9 °C, Grade 3: >= 39°C), headache, malaise, and myalgia (Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significant; prevents daily activity. Number of participants with any of the Grade (1, 2 or 3) and with each Grade (1, 2 and 3) solicited injection-site and systemic reactions were reported.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on Safety Analysis Set which included participants who have received at least one dose of the study vaccine and have any safety data available. Here 'number analyzed' signifies number of participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW Conjugate Vaccine | Menactra ®
Number analyzed (Participants) | 402 | 407
Participants
  Pain-Any Grade: number analyzed (Participants) | 398 | 402
  Pain-Any Grade | 178 | 196
  Pain-Grade 1: number analyzed (Participants) | 398 | 402
  Pain-Grade 1 | 141 | 154
  Pain-Grade 2: number analyzed (Participants) | 398 | 402
  Pain-Grade 2 | 33 | 34
  Pain-Grade 3: number analyzed (Participants) | 398 | 402
  Pain-Grade 3 | 4 | 8
  Erythema-Any Grade: number analyzed (Participants) | 398 | 402
  Erythema-Any Grade | 20 | 6
  Erythema-Grade 1: number analyzed (Participants) | 398 | 402
  Erythema-Grade 1 | 18 | 5
  Erythema-Grade 2: number analyzed (Participants) | 398 | 402
  Erythema-Grade 2 | 2 | 1
  Erythema-Grade 3: number analyzed (Participants) | 398 | 402
  Erythema-Grade 3 | 0 | 0
  Swelling-Any Grade: number analyzed (Participants) | 398 | 402
  Swelling-Any Grade | 16 | 3
  Swelling-Grade 1: number analyzed (Participants) | 398 | 402
  Swelling-Grade 1 | 13 | 1
  Swelling-Grade 2: number analyzed (Participants) | 398 | 402
  Swelling-Grade 2 | 3 | 2
  Swelling-Grade 3: number analyzed (Participants) | 398 | 402
  Swelling-Grade 3 | 0 | 0
  Fever-Any Grade: number analyzed (Participants) | 390 | 395
  Fever-Any Grade | 0 | 2
  Fever-Grade 1: number analyzed (Participants) | 390 | 395
  Fever-Grade 1 | 0 | 0
  Fever-Grade 2: number analyzed (Participants) | 390 | 395
  Fever-Grade 2 | 0 | 1
  Fever-Grade 3: number analyzed (Participants) | 390 | 395
  Fever-Grade 3 | 0 | 1
  Headache-Any Grade: number analyzed (Participants) | 398 | 402
  Headache-Any Grade | 151 | 134
  Headache-Grade 1: number analyzed (Participants) | 398 | 402
  Headache-Grade 1 | 90 | 73
  Headache-Grade 2: number analyzed (Participants) | 398 | 402
  Headache-Grade 2 | 52 | 47
  Headache-Grade 3: number analyzed (Participants) | 398 | 402
  Headache-Grade 3 | 9 | 14
  Malaise-Any Grade: number analyzed (Participants) | 398 | 402
  Malaise-Any Grade | 110 | 108
  Malaise-Grade 1: number analyzed (Participants) | 398 | 402
  Malaise-Grade 1 | 62 | 64
  Malaise-Grade 2: number analyzed (Participants) | 398 | 402
  Malaise-Grade 2 | 37 | 30
  Malaise-Grade 3: number analyzed (Participants) | 398 | 402
  Malaise-Grade 3 | 11 | 14
  Myalgia-Any Grade: number analyzed (Participants) | 398 | 402
  Myalgia-Any Grade | 146 | 156
  Myalgia-Grade 1: number analyzed (Participants) | 398 | 402
  Myalgia-Grade 1 | 98 | 120
  Myalgia-Grade 2: number analyzed (Participants) | 398 | 402
  Myalgia-Grade 2 | 40 | 27
  Myalgia-Grade 3: number analyzed (Participants) | 398 | 402
  Myalgia-Grade 3 | 8 | 9

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 up to Day 30 post-vaccination. Solicited Reaction (SR) were collected from Day 0 up to Day 7 post-vaccination.
Description: A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on Safety Analysis Set.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naive adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of a MenACYW Conjugate vaccine on Day 0.
- Group 2: Menactra ®: Healthy, meningococcal-vaccine naive adolescents (>= 15 to < 18 years) or adults (>= 18 years) received a single dose of Menactra vaccine on Day 0.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra ®
All-Cause Mortality (participants affected / at risk) | 0/402 | 0/407
Serious Adverse Events (participants affected / at risk) | 5/402 | 4/407
Other Adverse Events (participants affected / at risk) | 255/402 | 263/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=402) | Group 2: Menactra ® (N=407)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy To Arthropod Sting (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=402) | Group 2: Menactra ® (N=407)
Injection Site Pain (General disorders) | 178 (178) | 196 (196)
Malaise (General disorders) | 110 (110) | 108 (108)
Myalgia (Musculoskeletal and connective tissue disorders) | 147 (148) | 158 (161) — Myalgia events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Headache (Nervous system disorders) | 155 (168) | 137 (152) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.